CLINICAL TRIAL: NCT05040529
Title: Clinical Outcome of Living Donor Hepatectomy for Liver Transplantation: a Retrospective Study
Brief Title: Comparison Between Pure Laparoscopic Donor Right Hepatectomy and Convensional Donor Right Hepatectomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, JinHong Lim, Associate Professor, Gangnam Severance Hospital
Other Study IDs: 3-2021-0039
Record Dates: First submitted 2021-08-31; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Healthy Donors for Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PLDRH: patients who underwent pure laparoscopic donor right hepatectomy
  Interventions: Procedure: pure laparoscopic donor hepatectomy
- ODRH: patients who underwent conventaional open donor right hepatectomy
  Interventions: Procedure: conventional open donor hepatectomy

INTERVENTIONS:
Procedure: pure laparoscopic donor hepatectomy — pure laparoscopic donor hepatectomy: patients who underwent pure laparoscopic right or right extended hepatectomy for liver donation at gangnam severance hospital
  Groups: PLDRH
Procedure: conventional open donor hepatectomy — conventional open donor hepatectomy: patients who underwent conventional right or right extended hepatectomy for liver donation at gangnam severance hospital
  Groups: ODRH

SUMMARY:
Perioperative clincal outcome between PLDRH and conventional open donor right hepatectomy (ODRH) will be compared retrospectively.

DETAILED DESCRIPTION:
the superiority of laparoscopic liver resection was well known in terms of reduced blood loss and minimized hospital stay compared with open liver resection. However, pure laparoscopic donor hepatectomy is a challenging procedure for beginner liver surgeons because of the major vessel preservation required during liver parenchymal transection. this study was designed to identify the superiority of laparoscopic donor hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* patients received right or right extended hepatectomy for liver donation at gangnam severance hospital

Exclusion Criteria:

* none

Ages: 17 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A healthy person between the ages of 17 and 65 years who was willing to donate a liver was considered
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-03-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-03-28 (Estimated)

PRIMARY OUTCOMES:
blood loss during hepatectomy | intraoperative
  bleeding amount during hepatectomy will be calculated in mL. based on the blood in the sucker machine and the surgical towels.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Hong Lim, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severacne Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hong SK, Lee KW, Choi Y, Kim HS, Ahn SW, Yoon KC, Kim H, Yi NJ, Suh KS. Initial experience with purely laparoscopic living-donor right hepatectomy. Br J Surg. 2018 May;105(6):751-759. doi: 10.1002/bjs.10777. Epub 2018 Mar 26. PMID 29579333